CLINICAL TRIAL: NCT02053753
Title: A Double-Blind, Randomized, Single-Dose, Parallel-Group Study in Healthy Volunteers to Assess the Bioequivalence of a 120 mg Denosumab Subcutaneous Dose When Administered as Denosumab CP4 Drug Product or as Commercially Available Denosumab CP2 Drug Product
Brief Title: Bioequivalence Study of Denosumab CP4 Drug Product and Commercially Available Denosumab CP2 Drug Product
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20120186
Record Dates: First submitted 2014-01-31; First posted 2014-02-04 (Estimated); Results first posted 2017-12-29 (Actual); Last update posted 2017-12-29 (Actual); Status verified 2017-07

CONDITIONS: Healthy Volunteer
Keywords: denosumab, bioequivalence
MeSH Terms: interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug Product CP4 (Experimental): Participants received a single dose of 120 mg denosumab manufactured using the new CP4 process subcutaneously on day 1.
  Interventions: Drug: Denosumab CP4
- Drug Product CP2 (Experimental): Participants received a single dose of 120 mg denosumab manufactured using the current CP2 process subcutaneously on day 1.
  Interventions: Drug: Denosumab CP2

INTERVENTIONS:
Drug: Denosumab CP4 — Denosumab produced by a process referred to as CP4, administered subcutaneously.
  Arms: Drug Product CP4
Drug: Denosumab CP2 — Denosumab produced by a process referred to as CP2, administered subcutaneously.
  Other Names: XGEVA®
  Arms: Drug Product CP2

SUMMARY:
To evaluate the bioequivalence based on pharmacokinetics (PK) of a single 120 mg subcutaneous dose of denosumab administered to healthy volunteers using denosumab CP4 or denosumab CP2 drug products.

ELIGIBILITY:
Key Inclusion:

* Healthy male and female, ages ≥ 18 to ≤ 65 years (inclusive)
* Body weight > 60 to < 100 kg at time of screening
* Clinically acceptable physical exams and laboratory tests (blood hematology, blood chemistry, urinalysis) and no history or evidence of any clinically significant medical disorder that would pose a risk to subject safety or interfere with study evaluations or procedures
* Normal or clinically acceptable electrocardiogram (ECG) (12-lead reporting heart rate and PR, QRS, QT, and QTc intervals) at screening
* Willing to be confined to the research facility for 2 consecutive nights
* Subject will be available for follow-up assessments

Exclusion Criteria:

Prior diagnosis of bone disease, or any condition that will affect bone metabolism such as, but not limited to: osteoporosis, osteogenesis imperfecta, hyperparathyroidism, hyperthyroidism, hypothyroidism, osteomalacia, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, current flare-up of osteoarthritis and/or gout, active malignancy, renal disease (defined as glomerular filtration rate [GFR] < 45 mL/min), Paget's disease of the bone, recent bone fracture (within 6 months), malabsorption syndrome

* Presents with any psychiatric disorder, which may prevent the subject from completing the study or interfere with the interpretation of the study results
* Significant changes in physical activity during the 6 months before study drug administration or constant levels of intense physical exercise
* Prior use of any non-Amgen approved medications within 4 weeks or 5-half lives (whichever time period is longer) of study drug administration and for the duration of the study. This includes medications such as, but not limited to: bisphosphonates, fluoride, hormone replacement therapy (ie, estrogen) or selective estrogen receptor modulator, such as ralaxofene, calcitonin, strontium, parathyroid hormone or derivatives, supplemental vitamin D [>1000 IU/day], glucocorticosteroids, anabolic steroids, calcitriol, diuretics, over the counter medications, herbal supplements
* Positive for human immunodeficiency virus (HIV) at screening or known diagnosis of acquired immune deficiency syndrome (AIDS)
* Positive hepatitis B surface antigen (HepBsAg) (indicative of chronic hepatitis B) or detectable hepatitis C virus ribonucleic acid (RNA) by polymerase chain reaction (PCR) at screening (indicative of active hepatitis C - screening is generally done by hepatitis C antibody [HepCAb], followed by hepatitis C virus RNA by PCR if HepCAb is positive)
* Known sensitivity to any of the products to be administered during the study
* Prior denosumab administration
* Receiving or has received any investigational drug (or is currently using an investigational device) within 30 days before receiving study drug, or at least 10 times the respective elimination half-life (whichever period is longer) and for the duration of the study
* Women with a positive pregnancy test at screening or day-1
* Men and women of reproductive potential who are unwilling to practice a highly effective method of birth control while on study through 5 months after receiving the last dose of study drug. Highly effective methods of birth control include sexual abstinence (men, women); vasectomy; or a condom with spermicide (men) in combination with either barrier methods, hormonal birth control or intrauterine device (women)
* Women who are lactating/breastfeeding or who plan to breastfeed while on study through 5 half-lives after receiving the dose of study drug
* Women planning to become pregnant while on study through 5 months after receiving the dose of study drug
* Men with partners who are pregnant or planning to become pregnant while the subject is on study through 5 months after receiving the last dose of study drug
* Unwilling or unable to limit alcohol consumption throughout the course of the study. Alcohol is prohibited 24 hours prior to screening, 24 hours prior to check-in on day -1, and throughout confinement. Alcohol is also limited to no more than 2 drinks per day during the outpatient period of the study through completion of day 127 (EOS). A standard drink is equivalent to 12 ounces of regular beer, 8 to 9 ounces of malt liquor, 5 ounces of wine, or 1.5 ounces of 80 proof distilled spirits
* Positive urine screen for alcohol and/or drugs with a high potential for abuse at screening or day -1. Rescreening of the subject within 48 hours of a positive result is permitted
* Any other condition that might reduce the chance of obtaining data required by protocol or that might compromise the ability to give truly informed consent and/or comply with study procedures
* Osteonecrosis of the jaw (ONJ) or risk factors for ONJ such as invasive dental procedures (eg, tooth extraction, dental implants, oral surgery in the past 6 months), poor oral hygiene, periodontal, and/or pre-existing dental disease
* Recent tooth extraction (within 6 months of screening visit)
* Evidence of hypocalcemia at screening
* Known vitamin D deficiency
* Known intolerance to calcium or vitamin D supplements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2014-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (2):
- United States (2):
  - Research Site, Cypress, California
  - Research Site, San Antonio, Texas

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 2 centers in the United States.
Pre-assignment Details: Participants were randomized in a 1:1 ratio to receive a single 120-mg dose of denosumab either as a 1.7 mL single injection of 70 mg/mL denosumab produced using the new CP4 process or as a 1.7 mL single injection of 70 mg/mL denosumab produced from the current CP2 process.
Groups:
- Denosumab CP4: Participants received a single dose of 120 mg denosumab manufactured using the new CP4 process subcutaneously on day 1.
- Denosumab CP2: Participants received a single dose of 120 mg denosumab manufactured using the current CP2 process subcutaneously on day 1.
Period: Overall Study
Arm/Group | Denosumab CP4 | Denosumab CP2
Started | 72 | 74
Received Treatment | 71 | 71
Completed | 65 | 66
Not Completed | 7 | 8
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Decision by Sponsor | 1 | 1
Not completed — Lost to Follow-up | 4 | 3

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set defined as all participants who were enrolled and received denosumab.
Groups:
- Total: Total of all reporting groups
Arm/Group | Denosumab CP4 | Denosumab CP2 | Total
Number analyzed (Participants) | 71 | 71 | 142
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.9 (10.9) | 37.6 (11.3) | 38.3 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 33 | 62
  Male | 42 | 38 | 80
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 5 | 4 | 9
  Black (or African American) | 24 | 24 | 48
  Multiple | 3 | 1 | 4
  White | 39 | 42 | 81
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic/Latino | 20 | 23 | 43
  Not Hispanic/Latino | 51 | 48 | 99

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Drug Concentration (Cmax) of Denosumab
Description: Serum denosumab concentration-time data were analyzed by non-compartmental methods. Serum concentrations below the LLOQ (20.0 ng/mL) were set to 0 before data analysis.
Time Frame: Day 1 predose up to day 127
Population: The pharmacokinetic (PK) concentration analysis set includes all participants who received denosumab and had at least one PK sample collected. Two participants were excluded from all PK analyses because insufficient samples were available (≥ 3 missing consecutive samples) for calculation of PK variables.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Denosumab CP4 | Denosumab CP2
Number analyzed (Participants) | 71 | 69
μg/mL | 12.7 (3.53) | 11.8 (3.51)
Statistical Analysis 1: Comparison: Denosumab CP4 vs Denosumab CP2; Test type: Non-Inferiority or Equivalence — The 2 treatments were considered bioequivalent if the 90% CIs for the ratio of the geometric means were between 0.80 and 1.25; Ratio of Geometrc Means (CP4:CP2) = 1.084, 90% CI 2-sided [0.995 to 1.181] — The ratio and confidence interval of the geometric means are based on natural log scale data converted back to the original scale

2. Primary Outcome: Area Under the Drug Concentration-time Curve From Time 0 to 18 Weeks Post-dose (AUC0-18 Weeks) of Denosumab
Description: as for outcome 1
Time Frame: Day 1 predose up to day 127
Population: The PK concentration analysis set; 2 participants were excluded from all PK analyses because insufficient samples were available for calculation of PK variables and a further 11 participants were excluded from the analysis of AUC0-18 weeks because all samples after week 16 were missing.
Measure: Mean (Standard Deviation); unit: day*μg/mL
Arm/Group | Denosumab CP4 | Denosumab CP2
Number analyzed (Participants) | 64 | 65
day*μg/mL | 579 (190) | 555 (166)
Statistical Analysis 1: Comparison: Denosumab CP4 vs Denosumab CP2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Geometric Means (CP4:CP2) = 1.028, 90% CI 2-sided [0.934 to 1.131] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Time to Maximum Observed Concentration (Tmax) of Denosumab
Description: as for outcome 1
Time Frame: Day 1 predose up to day 127
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Denosumab CP4 | Denosumab CP2
Number analyzed (Participants) | 71 | 69
days | 6.9 [2.0 to 14] | 7.0 [3.0 to 21]

4. Secondary Outcome: Half-life (T1/2) of Denosumab
Description: as for outcome 1
Time Frame: Day 1 predose up to day 127
Population: The PK concentration analysis set; 2 participants were excluded from all PK analyses because insufficient samples were available for calculation of PK variables and a further 11 participants were excluded from the analysis of T1/2 because all samples after week 16 were missing.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Denosumab CP4 | Denosumab CP2
Number analyzed (Participants) | 64 | 65
days | 23.9 (10.1) | 22.4 (10.2)

5. Secondary Outcome: Area Under the Serum C-telopeptide (CTX1) Percent Inhibition-Time Curve From Time 0 to 18 Weeks Post-dose (AUEC0-18 Weeks)
Description: Serum CTX1 concentration-time data were analyzed by non-compartmental methods. Serum CTX1 concentrations below the LLOQ (0.0490 ng/mL) were set to 0.0490 ng/mL before data analysis.
  AUEC0-18 weeks was estimated using the linear-log trapezoidal method.
Time Frame: Day 1 predose up to day 127
Population: The pharmacodynamic (PD) analysis set includes all participants who received denosumab and had at least one sCTX1 sample collected.
  Eleven participants were excluded from the analysis of AUEC0-18 weeks because no samples after week 16 were collected.
Measure: Mean (Standard Deviation); unit: day*percent inhibition
Arm/Group | Denosumab CP4 | Denosumab CP2
Number analyzed (Participants) | 65 | 66
day*percent inhibition | 8380 (2050) | 8190 (2250)

6. Secondary Outcome: Maximum Percent Inhibition (Imax) of Serum CTX1
Description: Serum CTX1 concentration-time data were analyzed by non-compartmental methods. Serum CTX1 concentrations below the LLOQ (0.0490 ng/mL) were set to 0.0490 ng/mL before data analysis.
Time Frame: Day 1 predose up to day 127
Population: The pharmacodynamic analysis set includes all participants who received denosumab and had at least one sCTX1 sample collected.
Measure: Mean (Standard Deviation); unit: percent inhibition
Arm/Group | Denosumab CP4 | Denosumab CP2
Number analyzed (Participants) | 71 | 71
percent inhibition | 69.8 (17.0) | 70.3 (13.7)

7. Secondary Outcome: Time to Reach Maximum Percent Inhibition (Tmax) of Serum CTX1
Description: as for outcome 6
Time Frame: Day 1 predose up to day 127
Population: as for outcome 6
Measure: Median (Full Range); unit: days
Arm/Group | Denosumab CP4 | Denosumab CP2
Number analyzed (Participants) | 71 | 71
days | 3.01 [0.0 to 112] | 3.96 [1.0 to 126]

8. Secondary Outcome: Number of Participants With Adverse Events
Description: A treatment-related adverse event (TRAE) is any treatment-emergent adverse event (AE) that per investigator review has a reasonable possibility of being caused by the investigational product.
Time Frame: From the first dose of denosumab through day 126
Population: All participants who received denosumab
Measure: Number; unit: participants
Arm/Group | Denosumab CP4 | Denosumab CP2
Number analyzed (Participants) | 71 | 71
participants
  Any adverse event | 26 | 24
  Serious adverse events | 0 | 1
  AEs leading to discontinuation of denosumab | 0 | 0
  Fatal adverse events | 0 | 0
  Treatment-related adverse events (TRAEs) | 4 | 6
  Treatment-related serious adverse events | 0 | 0
  TRAEs leading to discontinuation of denosumab | 0 | 0
  Treatment-related fatal adverse events | 0 | 0

9. Secondary Outcome: Number of Participants Who Developed Anti-denosumab Antibodies
Time Frame: Predose on day 1, and days 29, 67 and 127
Population: All participants who received denosumab
Measure: Number; unit: participants
Arm/Group | Denosumab CP4 | Denosumab CP2
Number analyzed (Participants) | 71 | 71
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of denosumab through day 126
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Denosumab CP4 | Denosumab CP2
Serious Adverse Events (participants affected / at risk) | 0/71 | 1/71
Other Adverse Events (participants affected / at risk) | 26/71 | 24/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab CP4 (N=71) | Denosumab CP2 (N=71)
Abscess limb (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab CP4 (N=71) | Denosumab CP2 (N=71)
Goitre (Endocrine disorders) | 0 | 1
Eye pruritus (Eye disorders) | 1 | 0
Scleral discolouration (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gastric mucosa erythema (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Tooth loss (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Injection site reaction (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Vessel puncture site haematoma (General disorders) | 1 | 0
Vessel puncture site pain (General disorders) | 0 | 1
Conjunctivitis viral (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Pilonidal cyst (Infections and infestations) | 0 | 1
Pulpitis dental (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 2
Viral infection (Infections and infestations) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Tongue injury (Injury, poisoning and procedural complications) | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood calcium decreased (Investigations) | 2 | 2
Blood phosphorus decreased (Investigations) | 1 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 6 | 4
Haematuria (Renal and urinary disorders) | 0 | 1
Haematospermia (Reproductive system and breast disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.